CLINICAL TRIAL: NCT01512667
Title: A Single Dose Study to Investigate the Pharmacokinetics of Odanacatib (MK-0822) in Subjects With Renal Insufficiency
Brief Title: Pharmacokinetic Assessment of Single-Dose Odanacatib (MK-0822) in Subjects With Severe Renal Insufficiency (MK-0822-067)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0822-067
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — odanacatib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Severe Renal Insufficiency Group (Experimental): Single-dose administration of odanacatib 50 mg to participants with severe renal insufficiency.
  Interventions: Drug: MK-0822
- Healthy Matched Control Group (Experimental): Single-dose administration of odanacatib 50 mg to healthy matched control participants.
  Interventions: Drug: MK-0822

INTERVENTIONS:
Drug: MK-0822 — A single oral dose (50 mg tablet) of MK-0822 will be administered on Day 1 after an overnight fast.
  Other Names: odanacatib

SUMMARY:
This study will investigate and compare pharmacokinetics of a single 50 mg dose of odanacatib administered to participants with impaired renal/kidney function to those of a healthy matched control group. The primary hypothesis is that plasma AUC0-∞ of odanacatib in participants with impaired renal function is similar to that in matched healthy participants following a single 50 mg oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Not currently pregnant, nursing or planning to be pregnant through-out the course of the study; individual agrees to use specified contraception per protocol requirement for duration of study. Note: All females must have a serum pregnancy test to ensure and document negative test results prior to inclusion in the study.
* Body Mass Index (BMI) of up to 39.49kg/m^2
* Assessed to be in good health, including no clinically significant cardiac abnormalities based on results from an electrocardiogram (ECG) performed at pre-screening and/or prior to administration of study drug.
* Meets the requirements of the study in regard to current medication profile including: prescribed medications, caffeine, alcohol, over-the-counter drugs, herbals and nutritional products; with expected non-use of recreational (illicit) drugs associated with misuse, abuse and/or addiction.
* Agrees to adhere to all smoking and dietary restrictions associated with the study.
* Possess the ability to understand the study, grant voluntary informed consent, and willingly comply with all study requirements.

Inclusion Criterion Specific to Participants with Renal/Kidney Insufficiency:

* Creatinine clearance of <30 mL/min

Inclusion Criterion Specific to Healthy Volunteers:

* Creatine clearance of ≥ 90 mL/min (for healthy volunteers)

Exclusion Criteria:

* Does not meet the age requirement, is mentally or legally incapacitated, has or is expected to have significant emotional problems, and/or a history of a clinically significant psychiatric disorder.
* Diagnosed with a disease or medical condition which may pose a risk to the participant or may confound the study results.
* Has demonstrated or suspected stenosis (narrowing) of the renal artery, and/or has had a renal transplant and/or kidney removal.
* Has current, unstable, significant organ system disease(s) and/or cancer(s).
* Has had a surgical procedure, donated 1 unit of blood or received another investigational study medication within 4 weeks prior to the study's first dose of investigational product.
* Unable to refrain from or anticipates the use of any new medication, including prescription and non-prescription drugs and/or herbal remedies. Exceptions may include medications prescribed for prevention of disease or preservation of a healthy life.
* Uses any medication or agent that has the potential to significantly alter renal/kidney function.
* Unable to avoid taking diuretics (within 4 hours prior to and after dosing with the investigational product) or phosphate binders containing aluminum, calcium or lanthanum salts; iron supplements or other metal cations; antacids; or multivitamins containing iron or zinc (within 8 hours prior to dosing and 4 hours after dosing with the investigational product). Note: individuals prescribed to diuretics must be on a stable dose for at least 4 weeks prior to the study's start date in order to participate.
* History of multiple and/or severe allergies, has had a life-threatening reaction to a drug or other agent, and/or inability to tolerate prescription or nonprescription drugs and/or food.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2012-08-22 (Actual); Study Completion 2012-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Severe Renal Insufficiency Group | Healthy Matched Control Group
Started | 13 | 12
Matched Participants | 12 | 12
Unmatched Participants | 1 (Participant was not matched to a healthy control participant.) | 0
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Renal Insufficiency Group | Healthy Matched Control Group | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.9) | 55.6 (10.0) | 59.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of MK-0822 From Time 0 to Infinity (AUC0-∞) After Single Dose
Description: For healthy and severe renal insufficiency participants, plasma samples were collected from predose to 336 hours postdose for determination of AUC0-∞ (Total AUC). AUC0-∞ is a measure of total drug exposure.
Time Frame: Pre-dose and 1, 2, 4, 6, 9, 12, 16, 24, 32, 48, 72, 96, 120, 168, 240, and 336 hours postdose
Population: The per protocol population consisted of all matched participants who complied with the protocol sufficiently to ensure that results will likely exhibit the effects of treatment according to the underlying scientific model.
Measure: Least Squares Mean (95% Confidence Interval); unit: μM*hr
Arm/Group | Severe Renal Insufficiency Group | Healthy Matched Control Group
Number analyzed (Participants) | 12 | 12
μM*hr | 51.47 [38.96 to 67.99] | 32.12 [24.60 to 41.95]
Statistical Analysis 1: Comparison: Severe Renal Insufficiency Group vs Healthy Matched Control Group; Natural log-transformed plasma values were analyzed using an analysis of covariance (ANCOVA) model with a categorical factor for population (severe renal insufficiency participants, healthy matched control participants) and continuous covariates for age and body mass index (BMI). Data are back transformed to geometric least-squares mean ratio (GMR) (severe renal insufficiency / healthy) and 90% confidence intervals; Test type: Non-Inferiority or Equivalence — Similarity will be concluded if the GMR (severe renal insufficiency / healthy) is contained within the interval [0.40, 2.50]; GMR = 1.60, 90% CI 2-sided [1.15 to 2.23]

2. Secondary Outcome: Maximum Concentration (Cmax) of MK-0822 After Single Dose
Description: For healthy and severe renal insufficiency participants, plasma samples were collected from predose to 336 hours postdose for determination of Cmax.
Time Frame: Pre-dose and 1, 2, 4, 6, 9, 12, 16, 24, 32, 48, 72, 96, 120, 168, 240, and 336 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Severe Renal Insufficiency Group | Healthy Matched Control Group
Number analyzed (Participants) | 12 | 12
nM | 359.85 [300.29 to 431.22] | 246.09 [206.91 to 292.69]
Statistical Analysis 1: Comparison: Severe Renal Insufficiency Group vs Healthy Matched Control Group; Natural log-transformed plasma values were analyzed using an ANCOVA model with a categorical factor for population (severe renal insufficiency participants, healthy matched control participants) and continuous covariates for age and BMI. Data are back transformed to GMR (severe renal insufficiency / healthy) and 90% confidence intervals; Test type: Superiority or Other; GMR = 1.46, 90% CI 2-sided [1.18 to 1.81]

3. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-0822 After Single Dose
Description: For healthy and severe renal insufficiency participants, plasma samples were collected from predose to 336 hours postdose for determination of Tmax.
Time Frame: Pre-dose and 1, 2, 4, 6, 9, 12, 16, 24, 32, 48, 72, 96, 120, 168, 240, and 336 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Severe Renal Insufficiency Group | Healthy Matched Control Group
Number analyzed (Participants) | 12 | 12
hr | 18.01 [2.00 to 96.23] | 4.02 [2.00 to 96.00]

4. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MK-0822 After Single Dose
Description: For healthy and severe renal insufficiency participants, plasma samples were collected from predose to 336 hours postdose for determination of t1/2.
Time Frame: Pre-dose and 1, 2, 4, 6, 9, 12, 16, 24, 32, 48, 72, 96, 120, 168, 240, and 336 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Severe Renal Insufficiency Group | Healthy Matched Control Group
Number analyzed (Participants) | 12 | 12
hr | 73.9 (25.0) | 80.0 (20.7)

ADVERSE EVENTS:
Time Frame: Up to 15 days
Description: The safety population consisted of all participants who received at least one dose of the study drug.
Arm/Group | Severe Renal Insufficiency Group | Healthy Matched Control Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 6/13 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Renal Insufficiency Group (N=13) | Healthy Matched Control Group (N=12)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less